CLINICAL TRIAL: NCT04054115
Title: The Acute Effects of the Prostaglandin (Alprostadil) on Cerebral and Pulmonary Flow After the Bidirectional Cavopulmonary Connection
Brief Title: Acute Effects of the Prostaglandin (Alprostadil) on Cerebral and Pulmonary Flow
Acronym: Alprostadil
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Covid 19 and difficulty with recruitment
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Rajiv Chaturvedi, Staff Cardiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000060394
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Alprostadil; Injections

STUDY DESIGN:
Intervention Model Description: Patients with a bidirectional Glenn in their Pre-Fontan evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): 1. Baseline cardiac catheterization under GA. (Standard of Care, SOC)
  2. Transfer patient to MRI unit
  3. Baseline MRI
     1. Obtain ABG for pCO2 from existing femoral arterial access.
     2. Repeat pressure measurements with existing catheters at the SVC, RA and Aorta.
     3. MRI phase contrast imaging for flow measurements(SOC).
  4. During the MRI, Alprostadil infusion will be started and titrated to the target dose 0.1mcg/kg/min, provided there is a less than 20% drop in blood pressure from baseline.
  5. Post alprostadil infusion
     1. 1ml blood sample taken from existing femoral venous access for prostaglandin level.
     2. Repeat pressure measurements with existing catheters left at the SVC, RA and Aorta.
     3. Repeat MRI flow measurements
  7.Return to cath lab if further intervention required. 8.Recovery and monitoring for 4 to 6 hours prior to discharge(SOC).
  Interventions: Drug: Alprostadil 5 MCG Injection

INTERVENTIONS:
Drug: Alprostadil 5 MCG Injection — During the MRI, Alprostadil infusion will be started and titrated to the target dose, ensuring there is a less than 20% drop in blood pressure from baseline. Repeat pressure and MRI flow measurements once Alprostadil reaches 0.1mcg/kg/min.

SUMMARY:
The second stage operation towards single ventricle palliation is 'bidirectional cavopulmonary connection' (BCPC). The superior vena cava is connected to the pulmonary artery, diverting 'blue' blood from the upper body (including the brain) to the lungs. A successful BCPC requires sufficient and easy blood flow through the lungs. Alprostadil is the synthetic form of prostaglandin (hormone that causes dilation of blood vessels) and has been shown to increase blood flow in the brain hence increasing blood flow to the lungs after BCPC, potentially useful in managing children post BCPC with low flow to the lungs and thus poor oxygenation. This study propose to investigate acute effects of Alprostadil on different blood vessels after BCPC.

ELIGIBILITY:
Inclusion Criteria:• BCPC patients at time of routine pre-Fontan assessment: Cardiac catheterization and cardiac magnetic resonance imaging (CMR)

• Patients between the ages of 1 and 6 years old.

Exclusion Criteria:

* Patients who are hypersensitive to this product or to any ingredient in its formulation.
* Patients with seizure disorders or coagulopathies.
* Patients with abnormal kidney function.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | will be measured 30 minutes to 40 minutes after infusion of alprostadil
  Cerebral blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Chaturvedi, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada